CLINICAL TRIAL: NCT00917098
Title: Behavior Therapy for Pediatric Trichotillomania
Brief Title: Examining Behavior Therapy for Trichotillomania in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH077197 (NIH); R01MH077197 (NIH); DSIR 84-CTS
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Trichotillomania
Keywords: Behavior Therapy; Supportive Counseling; Child; Adolescent; Hair Pulling; CBT
MeSH Terms: conditions — Trichotillomania | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavior Therapy (Experimental): Participants will receive behavior therapy during Phases 1 and 2.
  Interventions: Behavioral: Behavior Therapy
- Supportive Counseling (Placebo Comparator): Participants will receive supportive counseling during Phase 1 and will not participate in Phase 2.
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Behavior Therapy — Eight weekly sessions during Phase 1 and four sessions every other week during Phase 2; participants will work on implementing habit reversal techniques with psychoeducation, cognitive restructuring, and relaxation, if necessary
  Arms: Behavior Therapy
Behavioral: Supportive Counseling — Eight weekly sessions during Phase 1 of psychoeducation, support, and emotion management related to trichotillomania and other stressors
  Arms: Supportive Counseling

SUMMARY:
This study will evaluate a treatment for trichotillomania, or compulsive hair pulling, in children and adolescents.

DETAILED DESCRIPTION:
Trichotillomania (TTM) is a chronic impulse control disorder that causes people to pull out their own hair. TTM typically develops in late childhood or early adolescence. It has been suggested that, like with obsessive-compulsive disorder, early identification and treatment of TTM might prevent the disorder and other co-occurring disorders in adults. The researchers in this study have developed the first treatment for TTM to target children and adolescents. Preliminary trials of this treatment, called behavior therapy (BT), indicate efficacy. This study is a larger, more rigorous examination of whether BT can successfully treat children and adolescents with TTM.

Participation in this study will be divided into two phases, each lasting 8 weeks. Follow-up visits will occur 3 and 6 months after completing treatment. In Phase 1, participants will be randomly assigned to receive either BT or supportive counseling (SC) for their TTM. Both groups of participants will complete eight weekly study visits. Those receiving BT will be encouraged to identify situations in which hair pulling is likely to occur and use behavioral techniques to resist urges to pull their hair. BT will also involve self-monitoring and homework throughout the week. Those receiving SC will discuss ways to minimize interference of hair pulling with everyday life and receive education and emotional support from a study therapist-but will not be taught specific behavioral techniques. After 8 weeks, participants will be evaluated to determine whether treatment is helping them. If participants are receiving BT and showing reduction in symptoms, they will continue to Phase 2, which involves four maintenance sessions of BT over 8 weeks. If participants receiving BT are not responding to treatment, they will be given referrals to other services. Participants receiving SC will end their participation after 8 weeks, and those not responding to treatment will be offered BT.

Study assessments will be completed at baseline, after Phase 1, after Phase 2, and at 3- and 6-month follow-ups. These assessments will include a clinical interview, questionnaires about symptoms, and family assessment measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or symptoms of trichotillomania
* Presence of stable parent or guardian

Exclusion Criteria:

* Presence of another primary or co-primary psychiatric disorder that requires initiation of different active current treatment
* Current use of psychotropic medication (participants may be able to stop taking medications to start with study)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2008-10; Primary Completion 2014-03-26 (Actual); Study Completion 2014-03-26 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale (CGIS) | Measured at baseline; Weeks 4, 8, 12, and 16; and 3- and 6-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Martin E. Franklin, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Child and Adolescent OCD, Tic, Trichotillomania, and Anxiety Group (COTTAGe), Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Click here for information about the University of Pennsylvania Child & Adolescent OCD, Tic, Trich, & Anxiety Group — http://www.med.upenn.edu/cottage/